CLINICAL TRIAL: NCT05956626
Title: A PHASE 1 STUDY TO ASSESS THE SAFETY AND EFFICACY OF OCU410ST FOR STARGARDT DISEASE AND PHASE 2/3 PIVOTAL CONFIRMATORY CLINICAL TRIAL TO ASSESS THE SAFETY AND EFFICACY OF OCU410ST FOR STARGARDT DISEASE
Brief Title: A Phase 2/3 Trial to Assess the Efficacy and Safety of OCU410ST for Stargardt Disease
Acronym: GARDian3
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ocugen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: OCU410ST-101/301; OCU410ST-101 (Other: Ocugen)
Record Dates: First submitted 2023-06-30; First posted 2023-07-21 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Stargardt Disease
Keywords: ABCA4-associated retinopathies
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two phases.
  Phase 2/3 Pivotal Confirmatory Clinical Trial is a randomized, outcome assessor-masked, multicenter study.
  A total of fifty-one (51) subjects will be enrolled in a 2:1 ratio to either the treatment group (n=34 subjects) or to an untreated control group (n=17 subjects).
  Treatment group: 34 subjects. Subjects will receive a single subretinal injection of 200 µL OCU410ST in concentration of 1.5×10E11 vg/mL.
  Control group: 17 subjects. Subjects who are enrolled in the untreated control group of the study will not receive any treatment. They will be followed according to the same treatment schedule as the treated subjects.
  Phase 1 was a multicenter, open-label, dose-ranging/dose escalation study. A 3+3 study design will be used for the sequential dose-escalation cohorts in which subjects will receive a single subretinal injection of OCU410ST. Enrollment is complete for Phase 1.
Who Masked: Outcomes Assessor
Masking Description: The masked biostatistician and other study team members identified by the masking plan
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 2/3 Randomized Treatment Arm (Experimental): Subjects will receive a single subretinal injection of 200uL OCU410ST in concentration of 1.5 x 10E11vg/mL
  Interventions: Drug: OCU410ST
- Phase 2/3 Randomized Control Arm (No Intervention): Subjects will not receive any active study intervention

INTERVENTIONS:
Drug: OCU410ST — Subretinal Administration of OCU410ST
  Arms: Phase 2/3 Randomized Treatment Arm

SUMMARY:
Phase 2/3 Pivotal Confirmatory Clinical Trial is a randomized, outcome assessor-masked, multicenter study, that will enroll fifty-one (51) subjects. Subjects will be enrolled in a 2:1 ratio to either the treatment group (n=34 subjects) or to an untreated control group (n=17 subjects).

Phase 1 is complete and closed for enrollment. It was a multicenter, open-label, dose ranging/dose escalation study that enrolled 9 subjects.

DETAILED DESCRIPTION:
Name of Investigational Product: OCU410ST Name of Active Ingredient: Adeno-associated viral vector 5 human RORA (AAV5-hRORA)

Title of Study: A PHASE 1 STUDY TO ASSESS THE SAFETY AND EFFICACY OF OCU410ST FOR STARGARDT DISEASE AND PHASE 2/3 PIVOTAL CONFIRMATORY CLINICAL TRIAL TO ASSESS THE SAFETY AND EFFICACY OF OCU410ST FOR STARGARDT DISEASE

Study Center(s): Approximately fifteen study centers in the US.

Background: Stargardt disease is an eye disease that causes vision loss in children and young adults. It is an inherited disease caused by faulty genes that cause buildup of fat deposits in the eye. Currently, there is no approved treatment available for Stargardt disease.

OCU410ST Product Information:

OCU410ST is an Adeno-Associated Virus serotype 5 containing human RORA for the treatment of Stargardt disease. Dysregulation in lipid metabolism, oxidative stress, and anti-inflammatory mechanisms are critical for pathogenesis and progression of Stargardt disease. The role of hRORA in regulating these gene pathways strongly suggests OCU410ST could restore homeostasis in the eye and thereby serve as a therapeutic candidate for Stargardt disease.

Phase 2/3 Pivotal Confirmatory Clinical Trial is a randomized, outcome assessor-masked, multicenter study.

A total of fifty-one (51) subjects will be enrolled in a 2:1 ratio to either the treatment group (n=34 subjects) or to an untreated control group (n=17 subjects).

Treatment group: 34 subjects. Subjects will receive a single subretinal injection of 200 µL OCU410ST in concentration of 1.5×10E11 vg/mL.

Control group: 17 subjects. Subjects who are enrolled in the untreated control group of the study will not receive any treatment. They will be followed according to the same treatment schedule as the treated subjects.

Note: Data will be collected for the untreated eye at Screening, 4-month, 8-month, 12-month, four (4) long-term safety follow-up visits, and early termination visit (if applicable).

Data will be collected for the treated eye at Screening, treatment Day 1, Day 2, Day 15, 4-month, 8-month, 12-month, four (4) long-term safety follow-up visits, and early termination visit (if applicable).

Enrollment in the Phase 1 study is complete. Phase 1 enrolled a total of nine subjects in low, medium and high dose cohorts.

Low Dose Cohort (3.75×10E10 vg/mL):

Three (3) Subjects received a single subretinal injection of 200 µL OCU410ST in low dose concentration (3.75×10E10 vg/mL).

Medium Dose Cohort (7.5×10E10 vg/mL):

Three (3) Subjects received a single subretinal injection of 200 µL OCU410ST in medium dose concentration (7.5×10E10 vg/mL).

High Dose Cohort (2.25×10E11 vg/mL):

Three (3) Subjects received a single subretinal injection of 200 µL OCU410ST in high dose concentration (2.25×10E11 vg/mL).

ELIGIBILITY:
Phase 2/3 Inclusion Criteria (applicable for both adult and pediatric subjects):

1. Males or females aged ≥5 years at the time of consent.
2. Subjects who have confirmed clinical and CLIA certified or equivalent genetic diagnosis of Stargardt disease (including ABCA4 related retinopathies).
3. Adult subjects who have BCVA of 75 letters or less in the study eye (20/32 Snellen equivalent) and Pediatric subjects who have a BCVA of 35 letters or better in the study eye (20/200 Snellen equivalent).
4. The study eye should have at least one well-demarcated area of atrophy with a minimum diameter of 300 microns, and total lesion size must add to less than or equal to ≤ 18 mm2 (approximately 7-disc areas).
5. Have detectable outer nuclear layer (ONL) in the macular region

Phase 2/3 Exclusion Criteria (applicable for both adult and pediatric subjects):

1. Participation in ongoing antiretroviral therapy treatment.
2. Participation in any experimental treatment or research study within 60 days before screening (any previous eye treatments involving gene therapy, stem cells, implanted retinal chips, injections into the eye, or participation in an Alkeus ALK-001 study within the past 6 months)
3. Macular atrophy secondary to any disease other than Stargardt Disease (STGD).
4. Presence of genetic mutations that mimic Stargardt Disease like ELOVL4, or PROM1.
5. Contraindication to subretinal injection or use of anesthesia (local and/or general).

Phase 1 was a multicenter, open-label, dose-ranging/dose escalation study. Enrollment is complete for Phase 1

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in atrophic lesion size as measured by Fundus Auto Fluorescence | 12 months (Screening to 12 months post OCU410ST administration)
  Change in the area of atrophy will be evaluated from the baseline measurements, using FAF to assess the loss of retinal layers.
Safety (Participants With Ocular and Non-ocular AEs (Adverse Events) and SAEs (Serious Adverse Events)) | 12 months (Screening to 12 months post OCU410ST administration)
  Safety will be determined by the number of ocular and non-ocular Study Drug-related adverse events (SDAE), treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Change from baseline in Low Luminance Visual Acuity (LLVA) | 12 months (Screening to 12 months post OCU410ST administration)
  Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Low Luminance Visual Acuity (LLVA) letter score. A higher score represents better vision.
Change from baseline in Best Corrected Visual Acuity (BCVA) | 12 months (Screening to 12 months post OCU410ST administration)
  Visual function of the study eye was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) letter score. A higher score represents better vision.

OTHER OUTCOMES:
Patients Global Impression of Change (PGIC) score | 12 months (Screening to 12 months post OCU410ST administration)
  The Patients Global Impression of Change (PGIC) score will be administered to the patients to assess the impact of treatment on quality of subject's life.
Care Giver Administered Global Impression of Change score | 12 months (Screening to 12 months post OCU410ST administration)
  The Caregiver Global Impression of Change (GIC) will be administered to caregivers to evaluate the impact of treatment on the patient's quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Murthy Chavali, MD, Ph.D., Study Director — Ocugen., Inc.
Locations (14):
- United States (14):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Consultants Medical Group, Sacramento, California
  - Vitreo Retinal Associates, P.A., Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Advanced Research, LLC, Pompano Beach, Florida
  - Retina Partners Midwest, P.C., Carmel, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Mississippi Retina Associates, Jackson, Mississippi
  - The Retina Institute, St Louis, Missouri
  - Duke Eye Center, Durham, North Carolina
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Valley Retina Institute, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No